CLINICAL TRIAL: NCT05217602
Title: Incentivizing Meditation App Habit Formation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Arizona State University (Other)
Collaborators: Calm.com, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: STUDY00014710
Record Dates: First submitted 2022-01-20; First posted 2022-02-01 (Actual); Last update posted 2022-11-22 (Actual); Status verified 2022-11

CONDITIONS: Stress; Adherence, Treatment
Keywords: Meditation; Anchoring; Mobile Application; Stress; Adherence Persistence; Rewards
MeSH Terms: conditions — Treatment Adherence and Compliance

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- AC+ARwdC (Experimental): Prescribed Calm usage = 10 minutes a day; Personalized anchoring plan for initiating any available meditation; Weekly text message reminders during the intervention period to reinforce the use of their anchoring plan; In-kind rewards only if they meditate using their anchoring plan on at least 8 days out of every 2 weeks (i.e., 14 days) during the 8 week intervention period (i.e., eligible for 4 prizes); $20 incentive for completing the baseline, week 8, and week 16 surveys
  Interventions: Behavioral: AC+ARwdC
- AC+RwdC (Experimental): Prescribed Calm usage = 10 minutes a day; Personalized anchoring plan for initiating any available meditation; Weekly text message reminders during the intervention period to reinforce the use of their anchoring plan; In-kind rewards if they meditate on at least 8 days out of every 2 weeks (i.e., 14 days) during the 8 week intervention period (i.e., eligible for 4 prizes); $20 incentive for completing the baseline, week 8, and week 16 surveys
  Interventions: Behavioral: AC+RwdC
- Usual Calm Control (UC) (Active Comparator): Prescribed Calm usage = 10 minutes a day; Personalized anchoring plan for initiating any available meditation; $20 incentive for completing the baseline, week 8, and week 16 surveys
  Interventions: Behavioral: Usual Calm Control (UC)

INTERVENTIONS:
Behavioral: AC+ARwdC — The Calm app is downloadable by participants onto their smartphone to access meditations and other Calm app features during the intervention period. Participants in the AC+ARwdC group will watch a video with information about the study, conditional rewards, and how to create an anchoring plan for their meditation habit. Weekly text message reminders will be sent during the intervention period to reinforce use of the anchoring plan. Participants in the AC+ARwdC group will be offered incentives for using their anchoring plan during the intervention period and for completing the baseline, post-intervention, and follow-up surveys.
  Arms: AC+ARwdC
Behavioral: AC+RwdC — The Calm app is downloadable by participants onto their smartphone to access meditations and other Calm app features during the intervention period. Participants in the AC+RwdC group will watch a video with information about the study, conditional rewards, and how to create an anchoring plan for their meditation habit. Weekly text message reminders will be sent during the intervention period to reinforce use of the anchoring plan. Participants in the AC+RwdC group will be offered incentives for meditating during the intervention period and for completing the baseline, post-intervention, and follow-up surveys.
  Arms: AC+RwdC
Behavioral: Usual Calm Control (UC) — The Calm app is downloadable by participants onto their smartphone to access meditations and other Calm app features during the intervention period. Participants in the UC group will watch a video with information about the study and how to create an anchoring plan for their meditation habit. Participants in the UC group will be offered incentives for completing the baseline, post-intervention, and follow-up surveys.
  Arms: Usual Calm Control (UC)

SUMMARY:
Over 75% of U.S. adults report significant stress, resulting in major health and economic costs. Mobile meditation apps are a feasible, effective, and scalable strategy for self-managing stress that is rapidly growing in popularity and thus represent a key tool for improving public health. However, existing intervention strategies for establishing persistent mobile health app adherence have largely been unsuccessful. Thus, there is a need for alternative strategies to move those who initiate meditation, i.e. new paying subscribers to a mobile meditation app. The investigators propose to synthesize theory- and evidence-based intervention approaches from psychology and behavioral economics to test novel combined strategies for establishing persistent adherence to meditation using the scalable Calm app.

The purpose of this study is to evaluate the use of anchoring strategies in combination with pragmatic in-kind rewards to identify the most optimal strategy for establishing persistent meditation habits with a mobile app. The investigators aim to assess the adherence persistence to a 10 minutes per day Calm prescription in new, paying self-initiated Calm subscribers; investigate the mediating effect of anchoring plan adherence on adherence persistence to the Calm prescription; and estimate the dynamic relationship between meditation adherence and stress. The investigators hypothesize that participants using anchoring strategies in combination with pragmatic in-kind rewards will be more likely to adhere to the Calm prescription than the control condition with greater adherence observed among those participating in the anchoring plus time-contingent reward intervention; greater adherence to anchoring plans will lead to higher adherence persistence; and greater reductions in stress will be associated with more persistent meditation adherence across study groups.

Investigators aim to recruit N=555 new, paying self-initiated Calm subscribers. Participants will be randomized into one of three groups with 185 participants in each group: anchoring plus in-kind rewards conditional on anchoring plan adherence; anchoring plus in-kind rewards conditional on meditating at any time of day; and usual Calm control condition without in-kind rewards.

DETAILED DESCRIPTION:
Stress among U.S. adults is widespread with major health and economic costs. Over 75% of U.S. adults report significant stress. Stress costs the U.S. $300 billion a year because of absenteeism, accidents, reduced productivity, employee turnover, and direct medical, legal, and insurance costs. There is an urgent need for accessible, effective, and scalable strategies to manage stress. This study employs an evidence-based mental health mobile app that is scalable.

Mobile meditation apps are a feasible, effective, and scalable strategy for self-managing stress that is rapidly growing in popularity and thus represent a key tool for improving public health. Given the ubiquity of smart phones, mobile health apps are an ideal platform for the remote delivery of health behavior regimens, such as meditation, as they can overcome several important barriers, such as cost and limited access, commonly reported by in-person programs. However, a majority of those who initiate use of a mobile meditation app do not persistently meditate and thus may not attain the corresponding mental health benefits. Recent research studies that have implemented app-based meditation have observed significant dropout and low adherence rates across different populations. Dropout rates have ranged from 54% to 77% among general samples of U.S. adults. Even when study participants do not officially drop out, adherence to app-based meditation interventions can be as low as 24%.

Existing intervention strategies for establishing persistent mobile health app adherence have largely been unsuccessful. Currently, little is known about how to get users to persistently adhere to a mobile health app. The significant rates of dropout and low adherence to mobile health apps indicate the presence of individual barriers to engagement. Proposed socio-cognitive intervention strategies have focused on bolstering self-efficacy for dealing with obstacles, increasing motivation, and reiterating the long-term benefits of performing a behavior, but to date, these strategies have largely been unsuccessful for establishing persistent health behaviors. Thus, there is a need for alternative strategies to move those who initiate meditation, i.e. new paying subscribers to a mobile meditation app, from preparation or action to maintenance. The investigators propose to synthesize theory- and evidence-based intervention approaches from psychology and behavioral economics to test novel combined strategies for establishing persistent adherence to meditation using the scalable Calm app.

Anchoring is a theory-based strategy for establishing persistent habits, but many participants need additional support to adhere to this approach. Psychologists have shown that repeatedly performing a behavior in response to the same stimulus or cue establishes a habit that can persist long term, i.e. beyond six months, with little or no cognitive effort. Through such "context-dependent repetition," exposure to the stimulus reflexively, or non-consciously, triggers initiation of the behavior. In this way, behavioral control is delegated to the external stimulus, thereby reducing the demand on an individual's attention and memory processes. Such external stimuli have been found to support many persistent health habits, such as high medication adherence, physical activity, reduced sitting, healthy hand washing, dental hygiene, and dietary habits.

Traditional external rewards that are unconditional on the timing and context of behavior can successfully initiate healthy behaviors, but the behaviors rarely persist after rewards are withdrawn. Behavioral economic theory predicts that short-term rewards will increase one's motivation to perform the targeted behavior and that short-term increases in behavioral performance increase one's utility or perceived benefit from continuing the behavior, thus forming a habit. The use of in-kind rewards, such as app-branded prizes like Calm merchandise, are often found to be more effective for increasing motivation than financial rewards. However, findings from the behavioral economics literature that used rewards, often financial incentives, show success only for initiating behavioral improvements across a wide range of health behaviors, such as physical activity, weight loss, and medication adherence, but a lack of success in maintaining the health behavior after rewards are withdrawn. Importantly, these studies all offered rewards for the targeted health behavior, unconditional on the timing and context of performing the behavior. Among the studies that evaluated the persistence of the health behavior after rewards were withdrawn, it is almost always found that the behavior returned to baseline levels of performance.

Time-contingent rewards may hold the key for leveraging the short-term effectiveness of rewards with the long-term efficacy of habits. One proposed explanation for the lack of long-term effectiveness of traditional rewards that are unconditional on the timing and context of behavior is that rewards crowd out motivation. However, one systematic review of health behavior interventions found that rewards increased health behavior motivation. One study found increased motivation from rewards for medication adherence, and also identified a subset for whom high medication adherence persisted after rewards were withdrawn: participants who used consistent stimuli or cues for their daily pill-taking. This observation, combined with the psychological theory of habits, informs the novel use of rewards conditional on anchoring plan performance for establishing persistent meditation adherence. One way to operationalize rewards for anchoring plan performance is to use "time-contingent" rewards that are conditional on performing the targeted behavior at approximately the same time that the planned anchor, i.e. existing routine, is expected to occur each day.

Therefore, the proposed intervention will test anchoring in combination with pragmatic in-kind rewards in two conditions: a) conditional on meditating at any time of day, and b) conditional on anchoring plan adherence, both compared to using Calm without additional strategies, to identify the most optimal strategy for establishing persistent meditation habits with a mobile app.

STUDY OBJECTIVES Aim 1: Assess adherence persistence to the 10 minutes per day Calm prescription in 555 new, paying self-initiated Calm subscribers for 16 weeks. H1.1: Over the 8-week follow-up period, participants in the intervention groups will be more likely to adhere to the 10 min/day Calm prescription than usual Calm condition. H1.2: Further, participants receiving pragmatic in-kind rewards tied to anchoring plan performance will have more persistent adherence than those receiving pragmatic in-kind rewards tied to meditation at any time of day.

Aim 2: Investigate the mediating effect of anchoring plan adherence during the 8-week intervention on adherence persistence to the Calm prescription. H2.1: Greater adherence to participants' anchoring plans during the intervention will lead to higher adherence persistence over the 8-week follow-up.

Aim 3: To estimate the dynamic relationship between meditation adherence and stress. H3.1: Greater reductions in stress will be associated with more persistent meditation adherence across study groups.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years of age
* New Calm subscribers (purchased at least 1 year membership)
* Able to read/understand English
* Have access to a smart phone on a daily basis
* Reside in the US or a US territory
* Willing to be randomized
* Have a Perceived Stress Scale score greater than or equal to 15

Exclusion Criteria:

* Greater than or equal to 60 minutes/month of meditation for the past six months

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 597 (Actual)
Dates: Start 2022-02-22 (Actual); Primary Completion 2022-10-31 (Actual); Study Completion 2022-10-31 (Actual)

PRIMARY OUTCOMES:
Mean Adherence Persistence Over Weeks 1-8 | Change from baseline to post-intervention (week 8)
  Mean Adherence Persistence over weeks 1-8 will be measured using Calm app usage data from weeks 1-8 of the study, retrieved from the Calm informatics team (with the participant permission). Mean adherence is measured as the percent of days per week with any meditation.
Mean Adherence Persistence Over Weeks 8-16 | Change from post-intervention (week 8) to follow-up (week 16)
  Mean Adherence Persistence over weeks 8-16 will be measured using Calm app usage data from weeks 8-16 of the study, retrieved from the Calm informatics team (with the participant permission). Mean adherence is measured as the percent of days per week with any meditation.

SECONDARY OUTCOMES:
Stress | Change from baseline to post-intervention (week 8) to follow-up (week 16)
  Stress will be measured using the Perceived Stress Scale. Scores on the PSS-10 range from 0-40 with greater scores indicating greater stress.
Anxiety | Change from baseline to post-intervention (week 8) to follow-up (week 16)
  Anxiety will be measured using the Hospital Anxiety and Depression Scale (Anxiety Subscale). Scores on the HADS Anxiety Subscale range from 0-21 with higher scores indicating greater anxiety.
Mindfulness | Change from baseline to post-intervention (week 8) to follow-up (week 16)
  Mindfulness will be measured using the Mindful Attention Awareness Scale. Scores on the MAAS range from 1-6 with higher scores indicating greater dispositional mindfulness.
PTSD | Change from baseline to post-intervention (week 8) to follow-up (week 16)
  PTSD will be measured using the Impact of Events Scale-Revised. Scores on the IES-R range from 0-88 with higher scores indicating greater severity of PTSD symptoms.
Sleep Disturbances | Change from baseline to post-intervention (week 8) to follow-up (week 16)
  Sleep Disturbances will be measured with the Insomnia Severity Index. Scores on the ISI range from 0-28 with higher score indicates more severe insomnia.
Habit Strength | Change from baseline to post-intervention (week 8) to follow-up (week 16)
  Habit Strength will be measured with the Self-Report Habit Index. Higher scores on the SRHI indicate greater habit strength.

CONTACTS AND LOCATIONS:
Overall Officials: Chad Stecher, PhD, Principal Investigator — Arizona State University
Locations (1):
- Arizona State University, Phoenix, Arizona, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Stecher C, Cloonan S, Linnemayr S, Huberty J. Combining Behavioral Economics-Based Incentives With the Anchoring Strategy: Protocol for a Randomized Controlled Trial. JMIR Res Protoc. 2023 Apr 28;12:e39930. doi: 10.2196/39930. PMID 37115610